CLINICAL TRIAL: NCT01582022
Title: The Effect of Bupivacaine (Marcaine) in Reducing Early Post Tonsillectomy Pain
Brief Title: Evaluation of The Effect of Bupivacaine (Marcaine) in Reducing Early Post Tonsillectomy Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Abdulmalik S. Alsaied, otolaryngology specialist, King Saud University
Allocation: Randomized | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-12-598
Record Dates: First submitted 2012-04-15; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Tonsillectomy
MeSH Terms: interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- local anesthetic (Experimental): local anesthetic agent
  Interventions: Drug: Bupivacaine
- normal saline (Placebo Comparator): comparator
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Bupivacaine — local application for 5 minutes
  Other Names: marcaine
  Arms: local anesthetic
Drug: normal saline — local application for 5 minutes
  Other Names: comparator
  Arms: normal saline

SUMMARY:
Research Methodology:

It will be a prospective, randomized, placebo-controlled, single-blind, intra-individual study in which one tonsillar fossa will be the tested side, and the other fossa will be the control. And the tested side will be packed with bupivacaine for five minutes. In the other hand, the controlled side will be packed for five minutes with gauze soaked in normal saline. The selection of the tested side and controlled side will be randomized based on the last digit in the medical record number (i.e. if the last digit is even then the tested side is the right and if the last digit is odd then the tested side is the left). Pain evaluation will be by visual analog scale and it will be in frequency of 2, 4, 6, 8, 12, 24 hours post-op.

DETAILED DESCRIPTION:
Evaluation of The Effect of Bupivacaine (marcaine) in Reducing Early Post Tonsillectomy Pain (Prospective, randomized, intra-individual study.) Study guidelines

Aim of the study

- to evaluate the effectiveness of applying bupivacaine intra-operative in reducing early post-tonsillectomy pain

Patients and methods

* It will be a randomized, placebo-controlled, single-blinded study
* one tonsillar fossa will be the tested side, and the other fossa will be the control
* to insure the random selection, the tested and control sides will be selected based on unpredicted method e.g. based on the last number in pt MRN: If the last # is even (0, 2, 4, 6, 8) = right side will be the tested If the last # is odd (1, 3, 5, 7, 9) = left side will be the tested
* Exclusion criteria included :

  1. pt with past history of unilateral peritonsillar abscess
  2. the current, regular use of a systemic steroid or NSAID
  3. a known hypersensitivity to bupivacaine
  4. a combined with unilateral myringotomy or bilateral myringotomy with unilateral ventilation tube
  5. pt with poor dental hygiene
* accompanied adenoidectomy is not an exclusion criteria
* the tested side will be : packed (after classic tonsillectomy) with gauze soaked in 0.5% bupivacaine, (2ml of bupivacaine + 2ml NS)for 5 min.
* the control side will undergoing the same of tested side but with normal saline
* post-operative analgesia will be paracetamol
* pain evaluation will be by visual analog scale (fig. 1) and it will be in frequency of 2, 4, 6, 8, 12, 24 hours post-op (frequency can be re-adjusted)
* Data of pain will be collected by the nurse. And they will not know which side is the tested. (single- blind)
* after phase I (data collection). Data will be calculated for P-value and other statistics scores
* Targeted sample size is 35 patients.
* patients will be consented for the possible adverse reactions of local application of the tested medicine (e.g. allergic reactions, Paresthesia). However, because in our study we will not add adrenaline, so differences in incidence of post-tonsillectomy bleeding is not expected.
* data will be statistically analyzed by McNemar's test
* For the data safety monitoring of the study, an independent external otolaryngology consultant (Dr.Ahmed Alarfij) will be assigned to monitor the safety of study participants.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing tonsillectomy

Exclusion Criteria:

1. pt with past history of unilateral peritonsillar abscess
2. the current, regular use of a systemic steroid or NSAID
3. a known hypersensitivity to bupivacaine
4. a combined with unilateral myringotomy or bilateral myringotomy with unilateral ventilation tube
5. pt with poor dental hygiene

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult